CLINICAL TRIAL: NCT04473963
Title: A Randomized Controlled Study to Evaluate the Reliability of Electrographic Flow™ (EGF) Mapping Algorithm Technology to Identify Sources of Atrial Fibrillation and Guide Ablation Therapy in Patients With Persistent Atrial Fibrillation
Brief Title: FLOW-AF: A Study to Evaluate Electrographic Flow™ (EGF) Mapping Technology
Acronym: FLOW-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cortex (Industry)
Collaborators: Ablacon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-001/002
Record Dates: First submitted 2020-03-16; First posted 2020-07-16 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation, Persistent
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Subjects will receive Electrographic Flow™ (EGF) mapping with Ablamap® Software. If EGF mapping identifies a source with a source activity level above threshold (≥26.5%) the subjects will be randomized to "treatment" or "control". If EGF mapping detects no source above threshold the subject will fall into the "not randomized" arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Randomized to Treatment: PVI + Electrographic Flow™ (EGF) Guided Ablation Therapy (Experimental): This arm includes subjects who underwent Electrographic Flow™ (EGF) mapping, and exhibited EGF-identified significant sources with leading source activity above threshold (≥26.5%), qualifying them for randomization.
  Subjects randomized to the "treatment" group first received pulmonary vein isolation (PVI) or PVI touch-up followed by a 20 minute waiting period and PVI confirmation. After this, EGF mapping in AF was conducted and targeted radiofrequency ablation of EGF-identified source(s) was performed in the left and right atrium. The procedure is considered complete once all EGF-identified sources have been eliminated through ablation. If necessary, the procedure were concluded with cardioversion.
  Interventions: Device: Electrographic Flow™ guided ablation
- Randomized to Control: PVI Only (No Intervention): This arm includes subjects who underwent Electrographic Flow™ (EGF) mapping, and exhibited EGF-identified significant sources with leading source activity above threshold (≥26.5%), qualifying them for randomization.
  Subjects randomized to the "control" group received standard pulmonary vein isolation (PVI) or PVI touch-up followed by a 20 minute waiting period and PVI confirmation. Subjects also received EGF mapping while in AF, but no further ablation of the EGF-identified sources. The procedure were concluded with cardioversion.
- Not Randomized (No Intervention): This arm includes subjects who underwent Electrographic Flow™ (EGF) mapping, but exhibited no EGF-identified sources with leading source activity above threshold (≥26.5%).
  Subjects received standard pulmonary vein isolation (PVI) or PVI touch-up followed by a 20 minute waiting period and PVI confirmation. Empiric adjunctive ablation could be performed at operator discretion. If necessary, the procedure were concluded with cardioversion.

INTERVENTIONS:
Device: Electrographic Flow™ guided ablation — In addition to standard pulmonary vein isolation (PVI) or PVI touch-up, subjects receive targeted radiofrequency source ablation guided by Electrographic Flow™ (EGF) mapping. EGF mapping enables the full spatiotemporal reconstruction of organized atrial electrical wavefront propagation to identify active sources or origins of excitation that may trigger atrial fibrillation (AF).
  EGF mapping involves 1 minute recordings of unipolar electrograms from a basket catheter, which are then processed with the EGF software. Several basket catheter positions are acquired in standard positions in both the left and right atria. EGF-identified sources with activity above the threshold (≥ 26.5%) are considered significant and targeted for ablation. The procedure concludes when all EGF-identified sources are eliminated, defined as reducing source activity below the threshold.
  Other Names: Electrographic Flow™ Mapping Technology; OptiMap™; Ablamap®
  Arms: Randomized to Treatment: PVI + Electrographic Flow™ (EGF) Guided Ablation Therapy

SUMMARY:
This study is to evaluate Electrographic Flow™ (EGF) mapping algorithm technology (Ablamap® Software).

DETAILED DESCRIPTION:
The objective of this study is to evaluate the reliability of Electrographic Flow™ (EGF) mapping algorithm technology (Ablamap® Software) to identify sources of atrial fibrillation and guide ablation therapy in patients with persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Suitable candidate for intra-cardiac mapping and ablation of atrial arrhythmias.
2. Above eighteen (18) years of age or of legal age to give informed consent specific to state and national law.
3. Subjects with a history of documented symptomatic, persistent or longstanding persistent atrial fibrillation < 36 months.
4. Subject agrees to comply with study procedures and be available (geographically stable) for follow-up visits for at least 12 months.
5. Treatment of atrial fibrillation with ablation therapy presenting with recurrent symptoms of atrial fibrillation (not applicable to De Novo subjects)

Exclusion Criteria:

1. Left atrial diameter > 5.5 cm.
2. Left ventricular ejection fraction (LVEF) < 35%.
3. Presence of intramural thrombus, tumor or abnormality that precludes vascular access, catheter introduction or manipulation.
4. Coagulopathy, bleeding diathesis or suspected procoagulant state.
5. Known allergies or intolerance to anticoagulant and antiplatelet therapies to be used in conjunction with the study or contrast sensitivity that cannot be adequately pre-treated prior to the ablation procedure.
6. Positive pregnancy test results for female patients of childbearing potential or breast feeding.
7. Acute or chronic medical condition that in the judgment of the investigator would increase risk to the patient or deem the patient inappropriate to participate in the study.
8. Mitral valve stenosis and/or severe mitral regurgitation.
9. Valvular atrial fibrillation.
10. Prosthetic valves.
11. New York Heart Association (NYHA) Class IV.
12. History of myocardial infarction (MI) within 3 months prior to procedure.
13. Atrial septal defect (ASD) or left atrial appendage (LAA) closure device.
14. Atrial fibrillation from a reversible cause (e.g., surgery, hyperthyroidism, sarcoidosis or pericarditis).
15. Life expectancy < 12 months based on medical history or the medical judgement of the investigator.
16. Presence of any transvenous pacing, Implantable cardioverter defibrillators (ICD), cardiac resynchronization therapy (CRT) leads.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, Principal Investigator — Principal Investigator - Czech Republic; Tamas Szili-Torok, MD, Principal Investigator — Principal Investigator - The Netherlands; Stefan Spitzer, MD, Principal Investigator — Principal Investigator - Germany
Locations (4):
- Nemocnice Na Homolce Hospital, Prague, Czech Republic, Czechia
- Germany (2):
  - Practice Clinic Heart And Vessels, Dresden, Saxony Land
  - University Heart and Vascular Center Hamburg, Hamburg
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reddy VY, Langbein A, Petru J, Szili-Torok T, Funasako M, Dinshaw L, Wijchers S, Rillig A, Spitzer SG, Bhagwandien R, Metzner A, Kong MH, Neuzil P. A Randomized Trial of Electrographic Flow-Guided Redo Ablation for Nonparoxysmal Atrial Fibrillation (FLOW-AF). JACC Clin Electrophysiol. 2024 Aug;10(8):1856-1869. doi: 10.1016/j.jacep.2024.03.040. Epub 2024 Jun 5. PMID 38842972
- [Derived] Kutinsky I, Nilsson KR, Mrlik M, Kong MH, Mehta N, Castellano S. Electrographic flow (EGF) mapping reveals sex-based differences in EGF patterns with women concentrated in phenotypes that benefit from EGF-guided ablation. J Interv Card Electrophysiol. 2026 Jan 7. doi: 10.1007/s10840-025-02184-8. Online ahead of print. PMID 41498861
- See also: A Randomized Trial of Electrographic Flow-Guided Redo Ablation for Nonparoxysmal Atrial Fibrillation (FLOW-AF) — https://doi.org/10.1016/j.jacep.2024.03.040

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 patients from the run-in cohort declined to return for protocol-mandated EGF re-mapping procedure after the initial blanking period.
Groups:
- Randomized to Treatment: PVI + Electrographic Flow™ (EGF) Guided Ablation Therapy: This arm includes subjects who underwent Electrographic Flow™ (EGF) mapping, and exhibited EGF-identified significant sources with leading source activity above threshold, qualifying them for randomization.
  Subjects randomized to the "treatment" group first received pulmonary vein isolation (PVI) or PVI touch-up followed by a 20 minute waiting period and PVI confirmation. After this, EGF mapping in AF was conducted and targeted radiofrequency ablation of EGF-identified source(s) was performed in the left and right atrium. The procedure is considered complete once all EGF-identified sources have been eliminated through ablation. If necessary, the procedure were concluded with cardioversion.
- Randomized to Control: PVI Only: This arm includes subjects who underwent Electrographic Flow™ (EGF) mapping, and exhibited EGF-identified significant sources with leading source activity above threshold, qualifying them for randomization.
  Subjects randomized to the "control" group received standard pulmonary vein isolation (PVI) or PVI touch-up followed by a 20 minute waiting period and PVI confirmation. Subjects also received EGF mapping while in AF, but no further ablation of the EGF-identified sources. The procedure were concluded with cardioversion.
- Not Randomized: This arm includes subjects who underwent Electrographic Flow™ (EGF) mapping, but exhibited no EGF-identified sources with leading source activity above threshold.
  Subjects received standard pulmonary vein isolation (PVI) or PVI touch-up followed by a 20 minute waiting period and PVI confirmation. Empiric adjunctive ablation could be performed at operator discretion. If necessary, the procedure were concluded with cardioversion.
Period: Overall Study
Arm/Group | Randomized to Treatment: PVI + Electrographic Flow™ (EGF) Guided Ablation Therapy | Randomized to Control: PVI Only | Not Randomized
Started | 22 | 24 | 34
Intention to Treat | 22 | 24 | 34
Per Protocol | 20 | 22 | 28
Per Protocol With Complete Follow-up (Including follow-up) | 19 | 21 | 28
Completed | 21 | 23 | 32
Not Completed | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Not inducible in AF | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intention to Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized to Treatment: PVI + Electrographic Flow™ (EGF) Guided Ablation Therapy | Randomized to Control: PVI Only | Not Randomized | Total
Number analyzed (Participants) | 22 | 24 | 34 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (9.5) | 69.1 (10.5) | 62.6 (7.3) | 65.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 10 | 28
  Male | 15 | 13 | 24 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 27.2 (4.3) | 29.3 (5.3) | 30.3 (4.2) | 29.1 (4.6)
Long-Standing Persistent Atrial Fibrillation [Count of Participants; unit: Participants] | 5 | 6 | 6 | 17
CHA2DS2-VASc score [Mean (Standard Deviation); unit: units on a scale [scale range: 0-9]] — Tool to describe risk of ischemic stroke in patients with AF. To help guide the decision to treat patients with anticoagulants. Calculated by adding the number of risk factors: Congestive Heart Failure, Hypertension, Age≥75, Diabetes, Stroke/TIA, Vascular Disease, Age 65-74 years and Female Sex. Each risk factor adds a point to the risk score, except for Age ≥ 75 years & Stroke/TIA, which both add 2 points. Score of 0 represents a patient having no additional risk factors. The ESC guidelines considers a score of 1 to be moderate risk and a score ≥ 2 to be high risk. Range: 0 (low) - 9 (high)
  units on a scale [scale range: 0-9] | 2.7 (1.5) | 3.1 (1.4) | 1.8 (1.0) | 2.4 (1.3)
LA Size (cm) [Mean (Standard Deviation); unit: cm] | 4.5 (0.5) | 4.4 (0.7) | 4.4 (0.5) | 4.4 (0.6)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: %] — Left ventricular ejection fraction (LVEF) is the central measure of left ventricular systolic function. LVEF is the fraction of chamber volume ejected in systole (stroke volume) in relation to the volume of the blood in the ventricle at the end of diastole (end-diastolic volume). Stroke volume (SV) is calculated as the difference between end-diastolic volume (EDV) and end-systolic volume (ESV). LVEF is calculated from:
  LVEF: [SV/EDV] x 100
  % | 56 (6) | 58 (6) | 56 (7) | 57 (6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Procedure Success
Description: Acute Procedure Success is defined as successful elimination of significant sources of electrographic flow (EGF) through targeted radiofrequency ablation. EGF-identified sources are significant when their leading source activity is above threshold. Successful elimination is defined as reduction of the source activity of the leading source below threshold upon post-ablation remapping using EGF mapping.
Time Frame: During the Procedure
Population: Per protocol population. Outcome Measure is only applicable to the group "Randomized to Treatment: PVI + EGF-Guided Ablation Therapy", because this outcome assesses the ability to eliminate EGF-identified sources through targeted source ablation. Other groups did not receive EGF-identified source ablation, and are therefore not included in analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized to Treatment: PVI + EGF Guided Ablation Therapy: This arm includes subjects who underwent Electrographic Flow™ (EGF) mapping, and exhibited EGF-identified significant sources with leading source activity above threshold (≥26.5%), qualifying them for randomization.
  Subjects randomized to the "treatment" group first received pulmonary vein isolation (PVI) or PVI touch-up followed by a 20 minute waiting period and PVI confirmation. After this, EGF mapping in AF was conducted and targeted radiofrequency ablation of EGF-identified source(s) was performed in the left and right atrium. The procedure is considered complete once all EGF-identified sources have been eliminated through ablation. If necessary, the procedure were concluded with cardioversion.
Arm/Group | Randomized to Treatment: PVI + EGF Guided Ablation Therapy
Number analyzed (Participants) | 20
Participants | 19

2. Primary Outcome: Number of Participants With Serious Adverse Events Related to the Procedure Through 7 Days
Description: Freedom from Serious Adverse Events (SAE) related to the procedure through 7 days following the index procedure.
Time Frame: 7 days
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Total: All Subjects in ITT population
Arm/Group | Randomized to Treatment: PVI + EGF Guided Ablation Therapy | Randomized to Control: PVI Only | Not Randomized | Total
Number analyzed (Participants) | 22 | 24 | 34 | 80
Participants | 0 | 0 | 2 | 2
Statistical Analysis 1: Comparison: Randomized to Treatment: PVI + EGF Guided Ablation Therapy vs Randomized to Control: PVI Only; Test type: Non-Inferiority — Non-inferiority between subjects Randomized to Treatment vs subjects Randomized to Control; p = 0.277, Chi-squared

3. Secondary Outcome: Number of Electrographic Flow™ (EGF) Identified Sources With Consistent Location Across Subsequent EGF-Guided Procedures
Description: This measure represents the number of Electrographic Flow™ (EGF) identified sources that remained consistent in anatomical location during subsequent EGF-guided procedures. The number and anatomical locations of EGF-identified sources for each subject were compared between the Index procedure and a subsequent EGF-guided procedure conducted ≥ 3 months later. A source was considered consistent if it was visible in the same anatomical location across both procedures.
Time Frame: Index Procedure until Recurrence Procedure
Population: A subgroup of 12 subjects (with a total of 18 Electrographic Flow™ (EGF) identified sources) from the "Randomized to Control," "Randomized to Treatment," or "Not Randomized" groups who returned for a subsequent EGF-guided procedure ≥ 3 months later. Consistency of these sources was evaluated before any randomization/treatment occurred, making inter-group comparisons inappropriate. Groups could be combined as the focus was on source consistency over time, not treatment assignment.
Measure: Number; unit: EGF-identified Sources
Units Other Than Participants: Sources above Threshold
Groups:
- Subset of Subjects Randomized to Control or Therapy: A subset of these patients that were randomized to control or treatment at index procedure and received a recurrence procedure ≥ 3 months after the index procedure, due to recurrence of atrial fibrillation (AF). In this recurrence procedure, EGF mapping was repeated and the anatomical location of the EGF-identified sources in the recurrence procedure were compared to those in the index procedure.
Arm/Group | Subset of Subjects Randomized to Control or Therapy
Number analyzed (Participants) | 12
Number analyzed (Sources above Threshold) | 18
EGF-identified Sources | 16

4. Secondary Outcome: Number of Participants With 12-month Freedom From AF Recurrence
Description: This measure represents the number of subjects with freedom from documented episodes of atrial fibrillation (AF) recurrence lasting longer than 30 seconds from the 90-day post-procedure blanking period through 12 months of follow-up. Follow-up and electrocardiographic monitoring of AF occurred at 3, 6 and 12 months through 7-day Holter recordings and ECGs.
Time Frame: 90 day - 12 months
Population: Per protocol population with completed 12 month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to Treatment: PVI + EGF Guided Ablation Therapy | Randomized to Control: PVI Only | Not Randomized
Number analyzed (Participants) | 19 | 21 | 28
Participants | 13 | 6 | 17
Statistical Analysis 1: Comparison: Randomized to Treatment: PVI + EGF Guided Ablation Therapy vs Randomized to Control: PVI Only; Test type: Equivalence — Equivalence between subjects "Randomized to Control" and subjects "Randomized to Treatment"; p = 0.042, Kaplan-Meyer Log Rank

5. Secondary Outcome: Average EGF Source Ablations Per Patient
Description: Average number of Electrographic Flow™ (EGF) source ablations per patients, defined as the number of significant EGF-identified sources with a source activity above threshold.
Time Frame: During the procedure
Population: Intention to Treat of the group "Randomized to Treatment"
Measure: Mean (Standard Deviation); unit: Source Ablations per Patient
Arm/Group | Randomized to Treatment: PVI + EGF Guided Ablation Therapy
Number analyzed (Participants) | 22
Source Ablations per Patient | 3.05 (1.89)

6. Secondary Outcome: Total Duration of EGF Source Ablation Per Patient
Description: Average total duration of radiofrequency ablation of the significant Electrographic Flow™ (EGF) identified sources per patient. Defined as the number of seconds of radiofrequency ablation spend on EGF-identified source ablation.
Time Frame: During the procedure
Population: Intention to Treat population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Randomized to Treatment: PVI + EGF Guided Ablation Therapy
Number analyzed (Participants) | 22
minutes | 10.18 (6.70)

7. Secondary Outcome: Average Fluoroscopy Time Per Patient
Description: Average total fluoroscopy time (in minutes) of the complete electrophysiology procedure per patient.
Time Frame: During the procedure
Population: Intention to Treat Population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Randomized to Treatment: PVI + EGF Guided Ablation Therapy | Randomized to Control: PVI Only | Not Randomized
Number analyzed (Participants) | 22 | 24 | 32
minutes | 15.1 (11.1) | 10.8 (7.2) | 13.8 (11.5)

8. Secondary Outcome: Total Radiation Dose Per Patient
Description: Average total radiation dose of the complete electrophysiology procedure, expressed in Air Kerma (AK) in mGy
Time Frame: During the procedure
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | Randomized to Treatment: PVI + EGF Guided Ablation Therapy | Randomized to Control: PVI Only | Not Randomized
Number analyzed (Participants) | 18 | 20 | 34
mGy | 155 (113) | 143 (151) | 186 (219)

9. Secondary Outcome: Total Procedure Time
Description: Total procedure time of complete electrophysiology procedure in minutes.
Time Frame: During the procedure
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Randomized to Treatment: PVI + EGF Guided Ablation Therapy | Randomized to Control: PVI Only | Not Randomized
Number analyzed (Participants) | 22 | 24 | 33
minutes | 183 (57) | 107 (34) | 137.2 (47)
Statistical Analysis 1: Comparison: Randomized to Treatment: PVI + EGF Guided Ablation Therapy vs Randomized to Control: PVI Only; Test type: Equivalence — Equivalence between procedure time of subjects "Randomized to Treatment" and subjects "Randomized to Control". The "Not-Randomized" group was not included in the analysis; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year follow-up after index procedure
Arm/Group | Randomized to Treatment: PVI + EGF Guided Ablation Therapy | Randomized to Control: PVI Only | Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24 | 2/34
Other Adverse Events (participants affected / at risk) | 3/22 | 3/24 | 5/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to Treatment: PVI + EGF Guided Ablation Therapy (N=22) | Randomized to Control: PVI Only (N=24) | Not Randomized (N=34)
Respiratory failure after presenting in volume overloaded state (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Respiratory failure after presenting in a volume overloaded state with acute decompensated heart failure. This event was adjudicated by an independend CEC as related to the procedure, but not related to the basket catheter or EGF mapping/ablation.
Arteriovenous fistula (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Right-sided arteriovenous fistula as a result of femoral venous access for the ablation procedure. This event was adjudicated by an independent CEC as related to the procedure, but not related to the basket catheter or EGF mapping/ablation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to Treatment: PVI + EGF Guided Ablation Therapy (N=22) | Randomized to Control: PVI Only (N=24) | Not Randomized (N=34)
Hematoma (Vascular disorders) | 3 (3) | 3 (3) | 5 (5) — Hematoma in groin. All of these were adjudicated by an independent CEC as related to the procedure, but not related to the basket catheter or EGF mapping/ablation.

LIMITATIONS AND CAVEATS:
The primary limitation of the FLOW-AF trial is the small number of patients enrolled. Although a statistically significant difference was seen between Electrographic Flow guided ablation vs the control condition, this trial was not powered to detect a difference between the treatment and control groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT04473963/Prot_SAP_000.pdf